CLINICAL TRIAL: NCT06618118
Title: A Phase 1 b Randomized, Double-blind, Placebo-Controlled, Experimental Medicine Study of Fosigotifator in Adults With Major Depressive Disorder
Brief Title: A Study to Assess Adverse Events of Fosigotifator (ABBV-CLS-7262) in Adults With Major Depressive Disorder
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-840; 2024-515120-36-00 (Other: EU CT)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder (MDD); Fosigotifator; ABBV-CLS-7262
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fosigotifator (Experimental): Participants will receive fosigotifator.
  Interventions: Drug: Fosigotifator
- Placebo (Placebo Comparator): Participants will receive matching placebo for fosigotifator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosigotifator — Oral Use
  Other Names: ABBV-CLS-7262
  Arms: Fosigotifator
Drug: Placebo — Oral Use
  Arms: Placebo

SUMMARY:
Major depressive disorder (MDD; depression) is a mood disorder that causes a continued feeling of sadness and loss of interest. It is a common and serious illness that can cause both emotional and physical symptoms such as feelings of sadness, irritability, not being able to focus on activities, tiredness, changes in eating habits, and aches and pains. The main goal of the study is to evaluate how safe and effective fosigotifator is in treating MDD.

Fosigotifator (ABBV-CLS-7262) is a new treatment being developed for adult patients with depression. This study is double-blinded, which means that neither the patients nor the study doctors know who is given fosigotifator and who is given placebo. Participants will be randomly assigned to one of the two groups to receive fosigatofator or placebo. There is 1 in 2 chance that participants will receive placebo. Approximately 106 adult participants with MDD will be enrolled in approximately 15 sites across the world.

Participants will receive oral fosigotifator or matching placebo. Duration of the study is approximately 144 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular weekly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 to 33 kg/m2 at the time of consent.
* Meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR) criteria for MDD based on the Structured Clinical Interview for DSM-5.
* Current major depressive episode of at least 6 weeks to less than 24 months in duration at Screening (Visit 1 ).
* Meets the following disease activity criteria mentioned in the protocol.
* Requires antidepressant therapy (ADT) per the investigator's opinion or, if currently taking ADT, must be able to safely discontinue ADT at least 7 days prior to the first dose of study drug at Baseline (Visit 2).

Exclusion Criteria:

- Primary psychiatric illness other than MDD.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 114 Days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - CenExel CNR /ID# 265866, Sherman Oaks, California
  - Clinical Neuroscience Solutions - Orlando - East South Street /ID# 265060, Orlando, Florida
  - CenExel iResearch, LLC /ID# 265886, Decatur, Georgia
  - Northwest Clinical Research Center /ID# 265057, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-840